CLINICAL TRIAL: NCT00005316
Title: White Coat Hypertension and Antihypertensive Treatment Effect - SCOR in Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4086; P50HL018323 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To investigate the mechanisms of white coat hypertension and study it further as a risk factor for heart damage.

DETAILED DESCRIPTION:
BACKGROUND:

The multidisciplinary SCOR examined causes, consequences, and treatments of human hypertension. A central theme was the renal basis for human hypertension. The subproject on white coat hypertension began in December of 1985.

DESIGN NARRATIVE:

In the longitudinal study, eighty patients with white coat hypertension were compared with 40 age- and sex-matched normotensives, and with 80 patients with sustained hypertension. The protocol consisted of (a) clinic blood pressure measurements made both by a physician and a nurse, (b) self-monitoring at home, (c) noninvasive ambulatory monitoring, (d) reactivity testing (cold pressor test, mental arithmetic, and isometric exercise) and (e) Korotkoff signal recording. Patients were also tested for early markers of disease (echocardiography and urine albumin).

The 80 patients in each of the two hypertensive groups were randomized to one of four treatment protocols (20 patients each); an alpha blocker, a beta blocker, a combined alpha- and beta-blocker, or an ACE inhibitor. The doses of medication were adjusted to produce similar reductions of clinic blood pressure in the different groups. The test battery (a-e) was reported during treatment.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-12; Study Completion 1995-11 (Actual)

REFERENCES:
- [Background] Liu JE, Roman MJ, Pini R, Schwartz JE, Pickering TG, Devereux RB. Cardiac and arterial target organ damage in adults with elevated ambulatory and normal office blood pressure. Ann Intern Med. 1999 Oct 19;131(8):564-72. doi: 10.7326/0003-4819-131-8-199910190-00003. PMID 10523216
- [Background] Cavallini MC, Roman MJ, Pickering TG, Schwartz JE, Pini R, Devereux RB. Is white coat hypertension associated with arterial disease or left ventricular hypertrophy? Hypertension. 1995 Sep;26(3):413-9. doi: 10.1161/01.hyp.26.3.413. PMID 7649575
- [Background] Pickering TG, Devereux RB, Gerin W, James GD, Pieper C, Schlussel YR, Schnall PL. The role of behavioral factors in white coat and sustained hypertension. J Hypertens Suppl. 1990 Dec;8(7):S141-7. PMID 2095382
- [Background] Pickering TG, James GD, Boddie C, Harshfield GA, Blank S, Laragh JH. How common is white coat hypertension? JAMA. 1988 Jan 8;259(2):225-8. PMID 3336140